CLINICAL TRIAL: NCT03964896
Title: Evaluating the Feasibility of a Nurse-Driven Telephone Triage Intervention for Cancer Patients Undergoing Chemotherapy in the Ambulatory Setting
Brief Title: Nurse-Driven Telephone Intervention in Improving Side Effects in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0300; NCI-2019-02651 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0300 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Breast Carcinoma; Head and Neck Carcinoma; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Sarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (telephone intervention) (Experimental): During standard of care chemotherapy, patients receive up to 18 telephone calls from a nurse using a standardized triage call script over 20 minutes.
  Interventions: Other: Survey; Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Survey — Complete survey
  Other Names: Survey Instrument
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone calls

SUMMARY:
This clinical trial studies how well a nurse-driven telephone intervention improves side effects in patients with cancer who are undergoing chemotherapy. Receiving calls from a nurse at home while receiving chemotherapy may improve the management of side effects and overall care in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the feasibility of a proactive nurse-driven telephone triage intervention for patients with cancer receiving first-line chemotherapy in the ambulatory setting.

SECONDARY OBJECTIVES:

I. To explore the symptom experience of patients receiving a nurse-driven telephone triage intervention while receiving chemotherapy in the ambulatory setting.

II. To explore the satisfaction of patients receiving a nurse-driven telephone triage intervention while receiving chemotherapy in the ambulatory setting.

III. To explore the frequency of emergency room visits and hospital admissions for symptom management by patients receiving a nurse-driven telephone triage intervention while receiving chemotherapy in the ambulatory setting.

OUTLINE:

During standard of care chemotherapy, patients receive up to 18 telephone calls from a nurse using a standardized triage call script over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Newly diagnosed patients with a breast, sarcoma, or head and neck cancer diagnosis preparing to undergo first-line, standard of care chemotherapy (patients with head and neck cancer may be undergoing concurrent first-line chemotherapy and radiation treatment)
* All chemotherapy treatment to be completed at the study institution

Exclusion Criteria:

* Patients who have received previous chemotherapy treatment for cancer
* Patients who will be receiving chemotherapy on research protocols
* Pregnant patients, as they may be on unique treatment protocols outside standard of care or have symptom needs that are beyond the scope of this intervention
* Patients who are unable to verbalize (e.g. due to tracheostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of completing nurse-driven telephone triage calls | Up to 25 weeks
  Completion is defined as the patient answering the call and completing the assessment; the target completion rate is set as 70%. Completion of nurse-driven calls will be assessed separately by center (breast, sarcoma, head and neck) and globally across all centers. The study will declare the intervention to be feasible within a center if the 90% confidence interval for completion rate is completely above 70% or contains 70%. To calculate the confidence interval, the study will construct a generalized linear mixed model with only a term for intercept.

SECONDARY OUTCOMES:
Symptom experience | Up to 25 weeks
  Will be measured using the MD Anderson Symptom Inventory (MDASI). This information will be summarized using graphical methods including box-plots and histograms, as well as summary statistics and 90% confidence intervals. The MDASI will be assessed by center and time point, as well as by time point across all centers.
Patient Satisfaction | Up to 25 weeks
  This information will be summarized using graphical methods including box-plots and histograms, as well as summary statistics and 90% confidence intervals. Satisfaction will be assessed by treatment group and by time point, as appropriate. They will also be assessed by center and again across all centers.
Number of emergency room visits | Up to 25 weeks
  This information will be summarized using graphical methods including box-plots and histograms, as well as summary statistics and 90% confidence intervals. Number of emergency room visits will be assessed by treatment group and by time point, as appropriate. They will also be assessed by center and again across all centers.
Number of hospital admissions | Up to 25 weeks
  This information will be summarized using graphical methods including box-plots and histograms, as well as summary statistics and 90% confidence intervals. Number of hospital admissions will be assessed by treatment group and by time point, as appropriate. They will also be assessed by center and again across all centers.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Jernigan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org